CLINICAL TRIAL: NCT07208500
Title: The Effect of Delayed Remote Ischemic Preconditioning on Postoperative Pulmonary Complications in Elderly Patients Undergoing Non-Cardiac Thoracic Surgery
Brief Title: Effect of Delayed Remote Ischemic Preconditioning on Postoperative Pulmonary Complications in Elderly Patients Having Non-Cardiac Thoracic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Geriatric Medical Center (Other)
Responsible Party: Principal Investigator, Xue Zhang, Attending Physician, Shanghai Geriatric Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B2025-038R
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Complications in Surgical Patients

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC Group (Experimental): Inflate a standard blood pressure cuff on one upper arm to 200 mmHg, maintain this pressure for 5 minutes, then deflate the cuff and keep it deflated for another 5 minutes. Repeat this process for 4 cycles.
  Interventions: Procedure: RIPC
- Control Group (Sham Comparator): Inflate a standard blood pressure cuff on one upper arm to 20 mmHg, maintain this pressure for 5 minutes, then deflate the cuff and keep it deflated for another 5 minutes. Repeat this process for 4 cycles.
  Interventions: Procedure: RIPC

INTERVENTIONS:
Procedure: RIPC — Inflate a standard blood pressure cuff on one upper arm to 200 mmHg, maintain this pressure for 5 minutes, then deflate the cuff and keep it deflated for another 5 minutes. Repeat this process for 4 cycles.

SUMMARY:
Study Summary: The Effect of a Simple Arm Cuff Procedure on Lung Complications After Surgery in Older Adults

1. What is the purpose of this study? This clinical study aims to find out if a simple, non-invasive procedure called Delayed Remote Ischemic Preconditioning (RIPC) can help reduce lung complications (like pneumonia or breathing difficulties) in older patients (aged 65 and above) after non-cardiac and non-chest surgery.
2. What is the RIPC procedure? RIPC involves briefly and repeatedly applying and releasing pressure on one upper arm using a standard blood pressure cuff. This is done 24 hours before surgery. The goal is to gently stimulate the arm's circulation, which may activate the body's natural protective mechanisms and help protect the lungs during and after surgery.

   RIPC Group: The cuff will inflate to a higher pressure (200 mmHg) for 5 minutes, then release for 5 minutes. This cycle repeats 4 times.

   Control Group: The cuff will inflate to a very low pressure (20 mmHg) with the same timing, serving as a comparison to see if the higher pressure has a specific effect.
3. Who can participate?

   Patients may be eligible if they:

   Are 65 years of age or older. Are scheduled for elective non-cardiac, non-chest surgery under general anesthesia, expected to last 1-3 hours.

   Are in relatively stable health (ASA physical status I-II). Patients cannot participate if they have certain pre-existing conditions, such as significant heart or lung disease, severe infections, or bleeding disorders.
4. What will happen during the study? Before Surgery: Eligible patients will receive a full explanation and sign a consent form. They will be randomly assigned (like flipping a coin) to either the RIPC group or the Control group. The procedure will be performed 24 hours before surgery. Some blood tests and an ultrasound scan will be done.

   During Surgery: Standard anesthesia and surgical care will be provided. After Surgery: We will monitor patients for any lung complications within 7 days after surgery. Additional blood tests and ultrasound scans will be performed to check lung function and look for signs of inflammation. We will also follow up 90 days after surgery to check on their overall recovery.
5. What are the potential benefits and risks? Potential Benefit: Participants may have a lower risk of developing postoperative lung complications. The knowledge gained may help future patients.

   Potential Risks: The arm cuff procedure may cause temporary discomfort, numbness, or minor bruising. There is a very small risk of more serious injury to the arm. The study team is trained to minimize these risks and will monitor patients closely. All standard risks associated with surgery and anesthesia still apply.
6. How is patient safety ensured? This study has been carefully reviewed and approved by an Ethics Committee to ensure it is scientifically sound and ethically conducted. Participation is voluntary, and patients can withdraw at any time without affecting their standard medical care. All personal information will be kept confidential. The study is sponsored and led by the Shanghai Geriatric Medical Center.

Study Version: V3.0 (September 2, 2025) Contact: For further questions, please contact the research team at the participating hospital.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients aged 65 years and above undergoing non-cardiac and non-thoracic surgery; operation time of 1-3 hours; American Society of Anesthesiologists (ASA) classification from I to II; BMI of 18-30 kg/m².

Exclusion Criteria:

* NYHA cardiac function classification is grade II to IV; there is severe respiratory dysfunction before surgery; there is a history of coagulation dysfunction diseases; chemotherapy, radiotherapy or immunotherapy have been received within 3 months; there is systemic or local active infection; there is peripheral vascular disease affecting upper limb blood vessels; antibiotics, non-steroidal anti-inflammatory drugs, or corticosteroids have been taken within the past 3 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of pulmonary complications 7 days after surgery | 7 days after surgery
  Postoperative pulmonary complications include: atelectasis, respiratory tract infection, respiratory failure, empyema, pulmonary embolism, bronchopleural fistula, and pneumothorax.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Geriatric Medical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No